CLINICAL TRIAL: NCT00548223
Title: Model Study on the Comprehensive Treating Protocol and Effect Evaluation of Ischemic Stroke With Traditional Chinese Medicine
Brief Title: The Secondary Prevention Trial for Ischemic Stroke With DengzhanShengmai Capsule
Acronym: SPIRITDZSM1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Nanhai Hospital of Traditional Chinese Medicine (Other); People's hospital of Huizhou city (Unknown); Taishan city hospital of TCM (Unknown); Ruijin Hospital (Other); First Affiliated Hospital of Fujian Medical University (Other); Yangjiang City Hospital of TCM in Guangdong Province (Unknown); Xinxing county hospital of TCM (Unknown); Southern branch of yuexiu district hospital of TCM (Unknown); Xinhui hospital of TCM of Jiangmen (Unknown); Shanghai Pudong New Area People's Hospital (Other); People's hospital of Jianyang city (Unknown); Luzhou Medical College (Other); Mianyang city hospital of TCM (Unknown); Guangyuan city hospital of TCM of Sichuan Province (Unknown); The Third Affiliated Hospital of Guangzhou Medical University (Other); Shunde district hospital of TCM (Unknown); Shenzhen People's Hospital (Other); Anyue County Hospital of Traditional Chinese (Other); Chengdu Integrated TCM&Western Medicine Hospital (Unknown); Guangzhou Red Cross Hospital (Other); Jiangsu Provincial People's Hospital (Other); Ankang Hospital of Traditional Chinese Medicine (Other); Qishan county hospital of shaanxi province (Unknown); Zongrui Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Lianyungang Chinese Medicine Hospital (Unknown); Yufu City Hospital of TCM in Guangdong Province (Unknown); 169 Military Hospital of China (Other); Affiliated Hospital of Liaoning University of Traditional Chinese Medicine (Other); The second affiliated hospital of shanxi college of TCM (Unknown); URUMQI Hospital of Traditional Chinese Medicine (Unknown); Hubei General Hospital (Unknown); The People's Hospital of Leshan (Other); Guagnzhou Liwan district Hospital of TCM (Unknown); Longhua Hospital (Other); Shanghai Jiao Tong University School of Medicine (Other); Hangzhou City Hospital of TCM (Unknown); Dongguan city hospital of TCM (Unknown); Liuzhou City hospital of TCM (Unknown); Maoming city hospital of TCM (Unknown); Beijing Tiantan Hospital (Other); Affiliated Hospital of Nantong University (Other); Xi'an city hospital of TCM (Unknown); Jiangsu province hospital of TCM (Unknown); The Third People's Hospital of Chengdu (Other); Huizhou Municipal Central Hospital (Other); Zhejiang Provincial Hospital of TCM (Other); The Second People's Hospital of Yibin (Other); Shanxi Provincial People's Hospital (Other Government); The First Affiliated Hospital of Guangzhou Medical University (Other); Guangxi Ruikang Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other); Afﬁliated Hospital of North Sichuan Medical College (Other); Third Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); ZhuHai Hospital (Other); Nanfang Hospital, Southern Medical University (Other); West China Hospital (Other); Guangdong Second Provincial Traditional Chinese Medicine Hospital (Industry); Handan First Hospital (Other); The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other); Conghua city hospital of TCM (Unknown); The First Affiliated Hospital of Guangxi University of Chinese Medicine (Unknown); Hubei Hospital of Traditional Chinese Medicine (Other); Jinan city hospital of TCM (Unknown); Shaanxi Hospital of Traditional Chinese Medicine (Other); Suining People's Hospital (Unknown); Wuzhou Red Cross Hospital (Other); Wuhan Interated ＆Western Hospital (Unknown); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Xi'an Central Hospital (Other); Zhengzhou City Hospital of Traditional Chinese Medicine (Other); Xiangya Hospital of Central South University (Other); Second Affiliated Hospital, Sun Yat-Sen University (Other); The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); ShuGuang Hospital (Other); Zhongshan Hospital Of Traditional Chinese Medicine (Other); Foshan Hospital of Traditional Chinese Medicine (Other); Teaching Hospital of Chengdu University of TCM (Unknown); Jiangmen Wuyi Hospital of Traditional Chinese Medicine (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, jianwen guo, MD, Professor, Guangzhou University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2006BAI04A02; 2006BAI04A02 (Other Grant/Funding Number: "Eleventh Five" program of China)
Record Dates: First submitted 2007-10-11; First posted 2007-10-23 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Stroke
Keywords: recurrence of stroke; Dengzhan Shengmai Capsule; Traditional Chinese Medicine
MeSH Terms: conditions — Stroke | interventions — dengzhan shengmai capsule

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dengzhan Shengmai capsule (Experimental): Dengzhan Shengmai capsule 0.18g by mouth twice a day for 1year
  Interventions: Drug: Dengzhan Shengmai capsule
- Placebo (Placebo Comparator): Placebo 0.18g by mouth twice a day for 1year
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dengzhan Shengmai capsule — Capsule, 0.18g, 2#, Bid*1year
  Other Names: DZSM
  Arms: Dengzhan Shengmai capsule
Drug: placebo — Capsule, 0.18g, 2#, Bid*1year
  Other Names: DZSMP
  Arms: Placebo

SUMMARY:
In order to observe the secondary preventive effect of the Dengzhanshengmai capsule on ischemic stroke, the investigators hold the large randomized control trial (RCT). 3143 subjects are included in 83 clinical research centers all over China. The subjects are randomly grouped into two groups. The basic therapy included antiplatelet aggregation, stroke health education, management of blood pressure, blood lipid and blood glucose, etc. The treating group will take the compound Chinese Medicine Deng Zhan Sheng Mai capsule and the contrast group will take the placebo for twelve months. Then all of the subjects are visited on the 30th, 90th, 180th, 360th day after inclusion. The recurrence of stroke, cardiovascular events, and peripheral arterial events are observed.

DETAILED DESCRIPTION:
Objective:To observe the secondary clinical effect of the Deng Zhan Sheng Mai capsule on ischemic stroke patients.

Methods:3143 subjects suffering from acute ischemic stroke are included in 83 clinical research centers all over China. The subjects are randomly divided into two groups:The treating group and the placebo group.Both groups accept the basic therapy and test drug.The basic therapy included antiplatelet aggregation,stroke health education,management of blood pressure,blood lipid and blood glucose,etc.The patients in Dengzhan Shengmaigroup take Deng Zhan Sheng Mai capsule and the placebo group take the placebo drug for twelve months.Then all of the subjects are visited on the 30th,90th,180th,360th day after inclusion. Primary endpoints(cerebral infarction,intracerebral hemorrhage,subarachnoid hemorrhage) and secondary endpoints(cardiovascular events,peripheral arterial disease),functional disability are observed at each follow up.

ELIGIBILITY:
Inclusion Criteria:

* 40-75 years old
* Ischemic stroke diagnosed by CT/MRI scan
* Patient presenting from 14 days to 6 months of first onset of ischemic stroke
* Presence of at least one risk factor of stroke (such as hypertension, diabetes mellitus, coronary heart disease, hyperlipidemia, and smoking, etc.) that can be interfered in
* Informed consent

Exclusion Criteria:

* Silent cerebral infarction
* Cerebral infarction due to other causes except artery scleroses (i.e. cardiogenic embolism, hypercoagulable state, endangium stripping, vasculitis)
* Presence of serious heart disease, heart, liver, lung, and kidney functional failure; malignancy; alimentary tract hemorrhage mental disorder and noncooperation with physician
* Females during pregnancy or lactation
* Already attend other clinical trial

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3143 (Actual)
Dates: Start 2007-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
recurrence of stroke | 1 year

SECONDARY OUTCOMES:
incidence rate of cardiovascular events, and peripheral arterial events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yan Huang, Bachelor, Principal Investigator — Guangdong Provincial Hospital of Tradtional Chinese Medicine
Locations (84):
- China (84):
  - Anhui College of Traditional Chinese Medicine First Affiliated Hospital, Hefei, Anhui
  - Xuanwu Hospital of Capital University of Medical Sciences, Beijing, Beijing Municipality
  - First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Dongguan City Chinese medicine hospital, Dongguan, Guangdong
  - Chinese medicine hospital in Foshan city, Foshan, Guangdong
  - Foshan First People's Hospital, Foshan, Guangdong
  - Integrated Hospital in Guangdong Province, Foshan, Guangdong
  - Foshan Shunde Area Integrated Hospital in Guangdong Province, Foshan, Guangdong
  - The second Chinese medicine hospital in Guangdong Province, Guangzhou, Guangdong
  - Guangdong Province Hospital of Tradtional Chinese Medicine, Guangzhou, Guangdong
  - Second Affiliated Hospital of Zhongshan University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong
  - Yuexiu area Hospital of TCM in Guangzhou, Guangzhou, Guangdong
  - Chinese medicine hospital in Liwan District of Guangzhou City, Guangzhou, Guangdong
  - Third Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong
  - Guangzhou Red Cross Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Third Affiliated Hospital of Zhongshan University, Guangzhou, Guangdong
  - People's Hospital of Huizhou City Center, Huizhou, Guangdong
  - Huizhou People Hospital in Guangdong Province, Huizhou, Guangdong
  - Jiangmen Wuyi Chinese medicine hospital, Jiangmen, Guangdong
  - Chinese medicine hospital Conghua City, Jiekou, Guangdong
  - Chinese medicine hospital in Maoming City, Maoming, Guangdong
  - Shenzhen City People's Hospital, Shenzhen, Guangdong
  - Taishan Hospital of TCM in Guangdong Province, Taishan, Guangdong
  - Xinhui Hospital of TCM in Guangdong Province, Xinhui District, Guangdong
  - Yangjiang Hospital of TCM in Guangdong Province, Yangjiang, Guangdong
  - Xinxing Hospitla of TCM in Guangdong Province, Yunfu, Guangdong
  - Chinese medicine hospital in Zhongshan City, Guangdong Province, Zhongshan, Guangdong
  - Chinese medicine hospital in Zhuhai, Guangdong Province Hospital, Zhuhai, Guangdong
  - Liuzhou Hospital of TCM in Guangxi, Liuchow, Guangxi
  - Ruikang Hospital Guangxi College of Traditional Chinese Medicine, Nanning, Guangxi
  - First Affiliated Hospital of Guangxi College of Traditional Chinese Medicine, Nanning, Guangxi
  - Guangxi Wuzhou Red Cross Hospital, Wuzhou, Guangxi
  - First Hospital of Handan City, Hebei Province, Handan, Hebei
  - The First Affiliated Hospital of Henan College of Traditional Chinese Medicine, Zhengzhou, Henan
  - Chinese medicine hospital in Zhengzhou City in Henan Province, Zhengzhou, Henan
  - Henan Province, the Third Affiliated Hospital of College of Traditional Chinese Medicine, Zhengzhou, Henan
  - Chinese medicine hospital in Hubei Province, Wuhan, Hubei
  - First Hospital of Wuhan City, Wuhan, Hubei
  - Wuhan University People's Hospital, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Hengyang Central Hospital, Hengyang, Hunan
  - The 169th Hospital of PLA, Hengyang, Hunan
  - Lianyungang Hospital of TCM in Jiangsu Province, Lianyungang, Jiangsu
  - Chinese medicine hospital in Jiangsu Province, Nanjing, Jiangsu
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangxi
  - Liaoning University of Traditional Chinese Medicine Affiliated Hospital, Shenyang, Liaoning
  - Chinese Medicine Hospital of Jinan City, Jinan, Shandong
  - Subsidiary of Shanghai University of Traditional Chinese Medicine, Longhua Hospital, Shanghai, Shanghai Municipality
  - Pudong New Area People Hospital in Shanghai, Shanghai, Shanghai Municipality
  - Ankang Hospital of TCM in Shanxi Province, Ankang, Shanxi
  - Qishan Hospital in Shanxi Province, Qishan, Shanxi
  - The 2nd affiliated Hospital fo Shanxi college of TCM, Taiyuan, Shanxi
  - Affiliated Hospital of Shaanxi College of Traditional Chinese Medicine, Xianyang, Shanxi
  - Chinese medicine hospital in Xi'an, Xi’an, Shanxi
  - Xi'an Central Hospital, Xi’an, Shanxi
  - Shaanxi Provincial People's Hospital, Xi’an, Shanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University Medical College, Xi’an, Shanxi
  - Chengdu Integrated Hospital, Chengdu, Sichuan
  - The Affiliated Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - People's Hospital of Sichuan Province, Chengdu, Sichuan
  - The 2nd People Hospital of Chengdu City, Chengdu, Sichuan
  - Guangyuan Hospital of TCM in Sichuan Province, Guangyuan, Sichuan
  - Jianyang Hospital of TCM in Sichuang Province, Jiancheng, Sichuan
  - Leshan City People's Hospital, Leshan, Sichuan
  - Affiliated Hospital of Luzhou Medical College, Luzhou, Sichuan
  - The Affiliated Hospital of TCM of Luzhou Medical School, Luzhou, Sichuan
  - Mianyang Hospital of TCM in Sichuan Province, Mianyang, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Anyue Hospital of TCM in Sichuan Province, Yueyang, Sichuan
  - Wulumuqi Hospital of TCM, Ürümqi, Xinjiang
  - Xinjiang Medical University Affiliated Hospital of First Clinical, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Zhejiang University of Traditional Chinese Medicine, Hangzhou, Zhejiang
  - Zhejiang University School of Medicine Second Affiliated Hospital, Hangzhou, Zhejiang
  - Chinese medicine hospital in Hangzhou, Hangzhou, Zhejiang
  - Ningbo City, Zhejiang Province zhongRui hospital, Ningbo, Zhejiang
  - Tiantan Hospital Capital University of Medical Sciences, Beijing
  - The Second Affiliated Hospital of Chongqing Third Military Medical University, Chongqing
  - Medical College of Shanghai Jiaotong University Yan Chai Hospital, Shanghai
  - Shanghai Jiaotong University Medical College Ruijin Hospital, Shanghai
  - Subsidiary of Shanghai University of Traditional Chinese Medicine ,Shuguang Hospital, Shanghai